CLINICAL TRIAL: NCT02891005
Title: A Multicenter, Prospective and Randomized Controlled Clinical Study (VasoguardTM Trial I) That Comparing the Safety and Efficacy of Paclitaxel Controlled Release Balloon Catheter (VasoguardTM) in the Treatment of Small Coronary Vessel Stenosis With a Common Coronary Balloon Catheter (Maverick2)
Brief Title: Comparing the Safety and Efficacy of Paclitaxel Controlled Release Balloon Catheter (VasoguardTM) in the Treatment of Small Coronary Vessel Stenosis With a Common Coronary Balloon Catheter (Maverick2)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Branden Med.Device Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Branden-123
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Small Vessel Lesion

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- paclitaxel controlled release balloon catheter (Experimental): Patients treated with paclitaxel controlled release balloon catheter
  Interventions: Device: paclitaxel controlled release balloon catheter (VasoguardTM)
- common balloon catheter (Experimental): Patients treated with common balloon catheter
  Interventions: Device: common balloon catheter (Maverick2)

INTERVENTIONS:
Device: paclitaxel controlled release balloon catheter (VasoguardTM) — paclitaxel controlled release balloon catheter implantation for small vessel lesion
  Arms: paclitaxel controlled release balloon catheter
Device: common balloon catheter (Maverick2) — common balloon catheter implantation for small vessel lesion
  Arms: common balloon catheter

SUMMARY:
Study Purpose The safety and efficacy of paclitaxel controlled release balloon catheter VasoguardTM in treatment of small vessel lesion.

Study Group Experimental group: paclitaxel controlled release balloon catheter (VasoguardTM) Control group: common balloon catheter (Maverick2)

ELIGIBILITY:
Inclusion Criteria:

Subject need 18 to 80 years of aged male or non-pregnant women; Subject has stable anina pectoris, or unstable anina pectoris, or old myocardial infarction patients, or ischemia with evidence but without symptom; Subject has a life expectancy of more than 2 years; Lesion vessel reference diameter is less than or equal to 2.5mm, target lesion length is less than or equal to 40mm; Target lesion stenosis is equal or greater than 70% or 50% and with ischemia; Single or two coronary small vessel lesions in situ; Subject can understand the trail purpose, sign informed consent voluntarily, agree to accept clinical telephone follow-up and angiographic follow-up at 9 months; Target lesion can be pre-expanded successfully (Guide wire can get through lesion, balloon pre-expand the remnant stenosis of vessel lumen is less or equal to 50%, without current limiting interlayer and thrombosis).

Exclusion Criteria:

Patient that in the opinion of the investigator is not appropriate for this trail; Pregnancy and lactation female patients; Patient has a life expectancy of less than 2 years; Severe congestive heart failure or NYHA IV heart failure; Patient who have bleeding constitution, cannot use antithrombotic and antiplatelet drugs; Patient that happened acute myocardial infarction within a week; Patient who happened stroke within six months; Patient who with severe renal failure (GFR≤30ml/Min); Patient has received heart transplantation; Patient who cannot tolerate aspirin and / or P2Y12 receptor inhibitor drugs; Patient who has allergy to paclitaxel, PLGA or contrast agent; Peptic ulcer or gastrointestinal bleeding within the prior 6 months; Patients who are participating in another drug or device clinical trail, which have not completed the primary endpoint follow- up period.

Angiographic relevant： Merge three or more coronary small vessel lesions; Target vessel with extensive thrombosis evidence; Restenosis of vein graft after bypass surgery; Target lesion proximal exist seriously distorted or severe calcified lesion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Late lumen loss | at 9 months

SECONDARY OUTCOMES:
Incidence of Device Success | at 9 months
Incidence of Operation Success | at 9 months
Incidence of the target lesion in-segment restenosis (%) at 9mm | at 9 months
Clinical-driven target lesion revascularization (TLR) and target vessel revascularization (TVR) | at 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Beijing, Beijing Municipality, China